CLINICAL TRIAL: NCT04255680
Title: A Study to Assess Variation in Potential Biomarkers in Friedreich Ataxia
Status: Completed | Type: Observational
Sponsor: Larimar Therapeutics, Inc. (Industry)
Collaborators: Children's Hospital of Philadelphia (Other)
Responsible Party: Sponsor
Other Study IDs: CLIN-1601-001
Record Dates: First submitted 2020-02-03; First posted 2020-02-05 (Actual); Last update posted 2020-08-18 (Actual); Status verified 2020-08

CONDITIONS: Friedreich Ataxia
MeSH Terms: conditions — Friedreich Ataxia | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Plasma, Buccal Cell and PAX Gene Blood Samples for RNA
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- FRDA Subjects: Male and female subjects with FRDA confirmed by genetic testing (aim for a 50:50 distribution of males to females)
  Interventions: Diagnostic Test: Buccal Swabs and Blood Draws
- Controlled Subjects: Male and female control subjects (matched by age [+/- 2 years] and sex)
  Interventions: Diagnostic Test: Buccal Swabs and Blood Draws

INTERVENTIONS:
Diagnostic Test: Buccal Swabs and Blood Draws — Buccal Swabs - Frataxin & specific RNA markers Blood Draws - Lipid panel, Uric Acid, Protein Marker Analysis and PAX Gene RNA Analysis

SUMMARY:
To test the variability of specific ribonucleic acid (RNA) and proteins as well as frataxin levels in samples of blood and buccal cells taken directly from patients with Friedreich's ataxia (FRDA) in order to confirm potential new biomarkers of disease in patients with FRDA.

DETAILED DESCRIPTION:
Primary Objective:

The primary objective of this study is to identify whether frataxin levels and specific RNAs and proteins in blood and buccal cells differ between patients with FRDA and controls.

Secondary Objective:

The secondary objectives of this study are:

* To understand the variability of frataxin and specific RNAs and proteins identified in buccal cells.
* To correlate levels of frataxin and specific RNAs and proteins with features of FRDA.
* To correlate levels of frataxin and specific RNAs and proteins with triglycerides, high density lipoprotein (HDL), low density lipoprotein (LDL) levels, and other lipids.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients with FRDA confirmed by genetic testing (FRDA subjects only).
2. Children and adults between the ages of 12 and 65 (inclusive); age for controls will be +/- 2 years relative to FRDA subjects.
3. Subject (and/or parent/legal guardian) has voluntarily signed consent form.
4. Willingness and ability to comply with all study procedures.
5. Functional Disability Stage (FDS) of 3, 4, or 5 (FRDA subjects only).

Exclusion Criteria:

1. Treatment with an investigational product within 30 days of study.
2. Use of gamma interferon or receiving any dose of gamma interferon within 90 days of the specimen collection day.
3. Use of any statin medications within 90 days of the specimen collection day.
4. Use of any lipid-lowering agents within 6 weeks of the specimen collection day.
5. Use of daily biotin supplementation that exceeds 30 mcg/day, either as part of a multivitamin or as a standalone supplement, within 7 days of the study visit.
6. Pregnant women.

Ages: 12 Years to 65 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: FRDA patients will be recruited using the Principal Investigator's (PI's) clinical practice.
  Control patients will be obtained through family members or friends of affected individuals, as well as non-FRDA patients in the PI's practice.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2020-01-14 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Difference in frataxin levels, specific RNAs and proteins | 1 day
  Difference in frataxin levels, specific RNAs and proteins between FRDA patients and control patients.

SECONDARY OUTCOMES:
Variability in frataxin levels, specific RNAs and proteins | 1 day
  Variability in frataxin levels, specific RNAs and proteins between FRDA patients and control patients.
Correlation of frataxin levels, specific RNAs and proteins in FRDA patients | 1 day
  Correlation of frataxin levels, specific RNAs and proteins with features of FRDA in patients with FRDA.
Correlation of frataxin levels, specific RNAs and proteins | 1 day
  Correlation of frataxin levels, specific RNAs and proteins with triglycerides, HDL, LDL and other lipid levels between FRDA patients and control patients.

CONTACTS AND LOCATIONS:
Overall Officials: David Lynch, M.D., Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Background] Coppola G, Burnett R, Perlman S, Versano R, Gao F, Plasterer H, Rai M, Sacca F, Filla A, Lynch DR, Rusche JR, Gottesfeld JM, Pandolfo M, Geschwind DH. A gene expression phenotype in lymphocytes from Friedreich ataxia patients. Ann Neurol. 2011 Nov;70(5):790-804. doi: 10.1002/ana.22526. PMID 22162061
- [Background] Coppola G, Marmolino D, Lu D, Wang Q, Cnop M, Rai M, Acquaviva F, Cocozza S, Pandolfo M, Geschwind DH. Functional genomic analysis of frataxin deficiency reveals tissue-specific alterations and identifies the PPARgamma pathway as a therapeutic target in Friedreich's ataxia. Hum Mol Genet. 2009 Jul 1;18(13):2452-61. doi: 10.1093/hmg/ddp183. Epub 2009 Apr 17. PMID 19376812